CLINICAL TRIAL: NCT00801528
Title: The Analgesic Efficacy of Continuous Wound Instillation With Diclofenac or Ropivacaine Following Cesarean Section: a Randomized, Double-blind, Placebo Controlled Study
Brief Title: Diclofenac vs. Ropivacaine for Cesarean Section
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Meir Medical Center (Other)
Responsible Party: Alex Khaikin MD, Meir Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MMC-0202-07
Record Dates: First submitted 2008-12-02; First posted 2008-12-03 (Estimated); Last update posted 2010-05-04 (Estimated); Status verified 2008-12

CONDITIONS: Cesarean Section
Keywords: ropivacaine; diclofenac; local anesthetic instillation
MeSH Terms: interventions — Ropivacaine; Diclofenac; Water; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Ropivacaine (Active Comparator): Continuous wound instillation of ropivacaine 0.2 % at a rate set of 10 mL/hr
  Interventions: Drug: Ropivacaine, Diclofenac, Water for injection
- Diclofenac (Active Comparator): Continuous wound instillation of diclofenac (300 mg/240 ml water for injection) at a rate set of 10 mL/hr
  Interventions: Drug: Ropivacaine, Diclofenac, Water for injection
- Water for injection (Placebo Comparator): Continuous wound instillation of water for injection at a rate set of 10 mL/hr
  Interventions: Drug: Ropivacaine, Diclofenac, Water for injection

INTERVENTIONS:
Drug: Ropivacaine, Diclofenac, Water for injection — Ropivacaine 0.2 %, or diclofenac (300 mg/240 ml water for injection) or water for injection will be administered as a constant instillation rate set of 10 mL/hr for the subsequent 18 postoperative hours.

SUMMARY:
A prospective, randomized, double blind study designed to investigate analgesic efficacy of wound infusion using diclofenac or ropivacaine following Cesarean section performed via a Pfannenstiel incision.

DETAILED DESCRIPTION:
Study Objective: To assess the analgesic efficacy of diclofenac or ropivacaine when administered via wound infusion.

Design: Prospective, randomized, double-blind, placebo-controlled study. Setting: Large referral hospital. Patients: 75 women recovering from Cesarean section performed via a Pfannenstiel incision.

Interventions: On completion of the surgical procedure, a 15 cm 19G infusion catheter (PAINfusor™, Baxter) will be placed below the fascia. According to a computer generated randomization schedule, patients will be divided into one of three treatment groups (n = 25).

* In Group Control water for injection will be administered.
* In Group Ropivacaine 0.2 % ropivacaine will be administered.
* In Group Diclofenac diclofenac (300 mg/240 ml of water for injection) will be administered.

During the first 6 postoperative hours, a co-investigator will administer "rescue" analgesia (10 ml bolus of infusion drug or rescue morphine). Thereafter, the catheter will be connected to an elastometric pump (LV 10 Infusor, Baxter) filled with either water for injection, ropivacaine 0.2 %, or diclofenac (300 mg/240 ml water for injection). The fluid will be administered as a constant infusion rate (10 mL/hr). Continuous wound infusion will be continued for the subsequent 18 postoperative hours. During this 18 hour period, subcutaneous morphine 4 mg will be administered on patient request for additional analgesia.

Measurements and Main Results: The following parameters will be assessed and recorded:

1. Demographic data
2. Surgical milestones(Anesthetic time, surgical time etc).
3. Incidence of failed intrathecal anesthesia
4. VAS for pain every 15 min during first 6 postoperative hours
5. Time to first pain (intrathecal anesthesia to VAS > 60 mm)
6. Number of infusion events (10 mL and 5 mL)
7. Rescue morphine administration during first 6 postoperative hours.
8. Subcutaneous morphine administration during subsequent 18 postoperative hours.
9. VAS for pain.
10. The incidence of nausea and vomiting.
11. Patient satisfaction at 24 hours, postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing Cesarean section

Exclusion Criteria:

A history of clinically significant disease:

* cardiovascular
* pulmonary
* hepatic
* renal
* neurologic
* psychiatric
* metabolic disease

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2008-04; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
1)Pain intensity 2)"Rescue" analgesia requirements | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Meir Medical Center, Kfar Saba, Israel